CLINICAL TRIAL: NCT02067065
Title: Non-anesthesiologist Administered Propofol Sedation for Colonoscopy - a Randomized Clinical Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Beatriz Ângelo (Other)
Responsible Party: Principal Investigator, Alexandre Ferreira, Dr, Hospital Beatriz Ângelo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: ColonPropo-01
Record Dates: First submitted 2014-02-16; First posted 2014-02-20 (Estimated); Last update posted 2015-10-12 (Estimated); Status verified 2015-10

CONDITIONS: Digestive System Diseases; Colonoscopy Sedation
Keywords: Colonoscopy; Sedation; Propofol; Non-anesthesiologist propofol administration
MeSH Terms: conditions — Digestive System Diseases | interventions — Colonoscopy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Non-anesthesiologist propofol sedation (Experimental): Bolus propofol sedation by non-anesthesiologist
  Interventions: Drug: Non-anesthesiologist propofol sedation; Procedure: Colonoscopy
- Anesthesiologist administered propofol (Active Comparator): Propofol sedation administered by an anesthesiologist
  Interventions: Drug: Propofol sedation administered by an anesthesiologist; Procedure: Colonoscopy

INTERVENTIONS:
Drug: Non-anesthesiologist propofol sedation — Bolus propofol sedation administered according to non-anesthesiologist propofol sedation guidelines of the European Society of Gastrointestinal Endoscopy
  Arms: Non-anesthesiologist propofol sedation
Drug: Propofol sedation administered by an anesthesiologist — Propofol sedation by an anesthesiologist
  Arms: Anesthesiologist administered propofol
Procedure: Colonoscopy — Elective total colonoscopy with or without biopsies, polypectomies or mucosal resection, as clinically indicated

SUMMARY:
Propofol is the preferred sedation for colonoscopy. There is debate on the safety of the administration of propofol by non-anesthesiologists, despite moderate quality evidence that support its' use.

There is only one small trial of a direct comparison of propofol sedation by anesthesiologists versus non-anesthesiologists.

Our aim is to compare the incidence of sedation related adverse events, the procedural quality indicators, times (onset, recovery, discharge) and patient satisfaction between non-anesthesiologist administered propofol sedation (NAAP) sedation and anesthesiologist propofol sedation.

A randomized clinical trial with the incidence of sedation related minor adverse events as primary endpoint will be conducted. Secondary endpoints include procedure quality indicators, propofol dosage and patient satisfaction.

A sample size of 330 subjects (2 arms of 165 patients) will be needed in order to obtain 90% power and a 5% significance level to exclude a 15% difference (15 - 30%) in adverse events incidence, estimated from our pilot experience. The sample size was adjusted for a 2% cross-over rate.

Informed and consenting patients undergoing colonoscopy examinations will be randomly assigned to one of two arms. One group will be sedated by an anesthesiologist according to a protocol of propofol mono-sedation. The other group will be sedated with propofol boluses, according to the European Society of Gastrointestinal Endoscopy (ESGE) NAAP guideline, with a 3-man team consisting of one endoscopist, one endoscopy nurse and a sedation nurse, trained in NAAP and exclusively dedicated to sedation and patient monitoring.

ELIGIBILITY:
Inclusion Criteria:

* Referred for elective colonoscopy as outpatients
* Must be able to provide the informed consent

Exclusion Criteria:

* American Society of Anaesthesiologists (ASA) class >2
* Pregnant women
* Difficult airway predictors (more than 2 ou Mallampati >3)
* Allergy to propofol or its' components
* IV drugs abuse

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 277 (Actual)
Dates: Start 2014-01; Primary Completion 2015-03 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Minor adverse events | During the sedation period
  Minor adverse events as defined by the International Sedation Task Force, including peripheral O2 saturation between 75-90% for less than 60 seconds, apnea, airway obstruction, sedation failure, allergic reaction without anaphylaxis, convulsion, brady/tachycardia and hypo/hypertension (>25% change from baseline)

SECONDARY OUTCOMES:
Propofol dosage | During the colonoscopy - an estimated mean time of 20 minutes
  Total propofol dosage
Patient satisfaction | Before discharge - estimated mean recovery time of 1 hour
  A 10 point visual scale on pain
colonoscopy quality indicators | During the procedure
  Colonoscopy quality indicators: time to cecum, withdrawal time, adenoma detection rate
Patient satisfaction 2 | Before discharge - estimated mean recovery time of 1 hour
  A 5 point likert scale on patient satisfaction with the sedation

CONTACTS AND LOCATIONS:
Overall Officials: Alexandre O Ferreira, MD, Principal Investigator — Hospital Beatriz Ângelo
Locations (1):
- Hospital Beatriz Ângelo, Loures, Portugal

REFERENCES:
- [Background] Dumonceau JM, Riphaus A, Aparicio JR, Beilenhoff U, Knape JT, Ortmann M, Paspatis G, Ponsioen CY, Racz I, Schreiber F, Vilmann P, Wehrmann T, Wientjes C, Walder B; NAAP Task Force Members. European Society of Gastrointestinal Endoscopy, European Society of Gastroenterology and Endoscopy Nurses and Associates, and the European Society of Anaesthesiology Guideline: Non-anesthesiologist administration of propofol for GI endoscopy. Endoscopy. 2010 Nov;42(11):960-74. doi: 10.1055/s-0030-1255728. Epub 2010 Nov 11. PMID 21072716
- [Background] Dumonceau JM, Riphaus A, Beilenhoff U, Vilmann P, Hornslet P, Aparicio JR, Dinis-Ribeiro M, Giostra E, Ortmann M, Knape JT, Ladas S, Paspatis G, Ponsioen CY, Racz I, Wehrmann T, Walder B. European curriculum for sedation training in gastrointestinal endoscopy: position statement of the European Society of Gastrointestinal Endoscopy (ESGE) and European Society of Gastroenterology and Endoscopy Nurses and Associates (ESGENA). Endoscopy. 2013 Jun;45(6):496-504. doi: 10.1055/s-0033-1344142. Epub 2013 May 23. No abstract available. PMID 23702777
- [Derived] Ferreira AO, Torres J, Barjas E, Nunes J, Gloria L, Ferreira R, Rocha M, Pereira S, Dias S, Santos AA, Cravo M. Non-anesthesiologist administration of propofol sedation for colonoscopy is safe in low risk patients: results of a noninferiority randomized controlled trial. Endoscopy. 2016 Aug;48(8):747-53. doi: 10.1055/s-0042-105560. Epub 2016 Apr 21. PMID 27100716